CLINICAL TRIAL: NCT01603277
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized Study to Evaluate the Safety, Tolerability, and Efficacy of KB003 in Subjects With Asthma Inadequately Controlled by Corticosteroids
Brief Title: Effect of KB003 in Subjects With Asthma Inadequately Controlled by Corticosteroids
Acronym: KB003-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB003-04
Record Dates: First submitted 2012-05-16; First posted 2012-05-22 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Moderate-to-Severe Asthma
Keywords: Asthma; GM-CSF; Moderate-to-Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-GM-CSF Monoclonal Antibody 400mg (Experimental)
  Interventions: Biological: Anti-GM-CSF Monoclonal Antibody 400mg
- Normal Saline (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Anti-GM-CSF Monoclonal Antibody 400mg — Anti-GM-CSF Monoclonal Antibody 400mg
  Arms: Anti-GM-CSF Monoclonal Antibody 400mg
Other: Placebo — Normal Saline
  Arms: Normal Saline

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of a single dose level of KB003 in subjects with inadequately controlled asthma.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of asthma established for at least 2 years
* Symptomatic asthma as defined by the Juniper Asthma Control Questionnaire
* Symptomatic asthma despite stable treatment with inhaled corticosteroids fluticasone or budesonide, or other corticosteroids, for at least 12 weeks
* Currently receiving inhaled long-acting beta agonist (LABA) or previously documented LABA intolerability or lack of responsiveness
* At least 2 exacerbations (no more than 6) in the previous 12 months that required systemic corticosteroids or at least a doubling of daily oral dose

Key Exclusion Criteria:

* Acute asthma worsening (requiring emergency room visit, hospitalization, urgent care, physician visit, or change in asthma medications) or lower respiratory tract infection requiring the use of antibiotics, within 4 weeks prior to Screening Visit.
* History of life-threatening asthma with admission to the intensive care unit requiring the use of mechanical ventilation within the past 12 months
* Use of any immunosuppressive or immunomodulatory agents within 12 weeks or an investigational agent within 4 weeks prior to Screening Visit
* History of any cardiovascular, neurological, hepatic, or renal condition
* History of smoking within the past 12 months

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor A. Molfino, MD, MSc, Study Chair — KaloBios Pharmaceuticals, Inc.
Locations (66):
- United States (30):
  - Birmingham, Alabama
  - Fullerton, California
  - Granada Hills, California
  - Los Angeles, California
  - Rancho Mirage, California
  - Sacramento, California
  - San Jose, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Waterbury, Connecticut
  - Miami, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Duluth, Georgia
  - Lawrenceville, Georgia
  - Savannah, Georgia
  - Lexington, Kentucky
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Reno, Nevada
  - Summit, New Jersey
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Arlington, Texas
  - Sugarland, Texas
  - Milwaukee, Wisconsin
- Australia (8):
  - Cairns, Queensland
  - Woolonggabba, Queensland
  - Bedford Park, South Australia
  - Woodville, South Australia
  - Box Hill, Victoria
  - Frankston, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- France (5):
  - Marseille
  - Montpellier
  - Rennes
  - Strasbourg
  - Tours
- Poland (9):
  - Bialystok, Podlaskie Voivodeship
  - Mrozy, Silesian Voivodeship
  - Wiłomin, Slaski
  - Biała Rawska
  - Bydgoszcz
  - Krakow
  - Lodz
  - Lublin
  - Piasta
- Ukraine (9):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Simferopol
  - Vinnytsia
  - Yalta
  - Zaporizhzhya
- United Kingdom (5):
  - Wishaw, Lanarkshire
  - Northwood, Middlesex
  - Bradford, West Yorkshire
  - Leeds, West Yorkshire
  - Southampton

REFERENCES:
- [Derived] Molfino NA, Kuna P, Leff JA, Oh CK, Singh D, Chernow M, Sutton B, Yarranton G. Phase 2, randomised placebo-controlled trial to evaluate the efficacy and safety of an anti-GM-CSF antibody (KB003) in patients with inadequately controlled asthma. BMJ Open. 2016 Jan 6;6(1):e007709. doi: 10.1136/bmjopen-2015-007709. PMID 26739717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 July 2012 - 09 June 2013
Period: Overall Study
Arm/Group | Anti-GM-CSF Monoclonal Antibody 400mg | Normal Saline
Started | 78 | 82
Completed | 64 | 64
Not Completed | 14 | 18
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 6 | 10
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Non-Compliance | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-GM-CSF Monoclonal Antibody 400mg | Normal Saline | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (11.95) | 53.1 (10.30) | 52.9 (11.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 73 | 135
  >=65 years | 16 | 9 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 34 | 34 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 69 | 69 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 74 | 75 | 149
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 59
  Poland | 26 | 19 | 45
  Ukraine | 17 | 17 | 34
  Australia | 6 | 7 | 13
  France | 1 | 4 | 5
  United Kingdom | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Predicted FEV1 at Week 24
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Anti-GM-CSF Monoclonal Antibody 400mg | Normal Saline
Number analyzed (Participants) | 78 | 82
Percent | 3.631 (12.6174) | 2.000 (8.5251)

2. Secondary Outcome: To Evaluate the Efficacy of KB003 as Measured by Asthma Exacerbation Rate
Time Frame: Week 24
Reporting Status: Not Posted

3. Secondary Outcome: To Evaluate the Effect of KB003 on Peak Expiratory Flow (PEF)
Time Frame: Week 24
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate the Safety and Tolerability of KB003 as Measured by Frequency and Severity of AEs, Clinical Safety, Laboratory Abnormalities and Chest Radiographic Assessments
Time Frame: Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Event Greater than or Equal to 5%
Arm/Group | Anti-GM-CSF Monoclonal Antibody 400mg | Normal Saline
Serious Adverse Events (participants affected / at risk) | 5/78 | 2/82
Other Adverse Events (participants affected / at risk) | 10/78 | 15/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-GM-CSF Monoclonal Antibody 400mg (N=78) | Normal Saline (N=82)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-GM-CSF Monoclonal Antibody 400mg (N=78) | Normal Saline (N=82)
Nasopharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Headache (Nervous system disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No